CLINICAL TRIAL: NCT04769154
Title: Adult Airway Management in The Intensive Care Units and Regular Floors: A Prospective Observational Study in A Tertiary Care Center
Brief Title: Adult Airway Management in the Intensive Care Units and Regular Floors
Status: Completed | Type: Observational
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Marie Awad, Professor and Chairperson, American University of Beirut Medical Center
Other Study IDs: BIO-2020-0049
Record Dates: First submitted 2021-02-23; First posted 2021-02-24 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Airway Management; Intensive Care Unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective observational study is to assess investigate the incidence of first attempt success rate of endotracheal intubation. Secondary objectives included assessing the predictors of first attempt success rate and the incidence and predictors of adverse events. The main question it aims to answer is whether endotracheal intubation outside the OR at AUBMC has higher success rates and lower complication rates as compared to the literature. Participants will be evaluated according to the inclusion criteria and data extraction will be performed from the electronic health record (EHR). Researchers will compare success and complication rates with previous literature and international benchmarks.

DETAILED DESCRIPTION:
Airway management is one of the pivotal roles of anesthesiologists that extends beyond the OR to include ICUs and regular hospital floors. Managing airways outside the OR is inherently complex and challenging. Numerous guidelines for non-OR airway management exist to assist practitioners. The American University of Beirut Medical Center (AUBMC), a tertiary care facility in a lower-to-middle-income country, experienced significant variation in practices concerning non-OR airway management, similar to other institutions. Nearly a decade ago, the quality, accreditation, and risk management department partnered with the Anesthesiology and Pain Management department to implement a care bundle for airway management outside the OR, excluding the Emergency Department (ED). This multidisciplinary approach prompted an assessment of our practices, aiming to compare our success and complication rates with the literature and international benchmarks.

This is a prospective observational study to evaluate the outcomes of endotracheal intubations for critically ill patients in ICUs and on regular floors. Data were prospectively collected by the anesthesia nurse assisting in the procedure or extracted from the electronic record as appropriate.

The sample size was calculated using the estimation of a simple proportion method (https://epitools.ausvet.com.au/oneproportion). Studies have shown a first attempt success rate of 75%. Based on these results, a sample size of 100 patients was calculated, based on an estimated proportion of 70%, a desired precision of estimate of 10%, a confidence level of 95%, and an estimated dropout rate of 20%. However, to improve the power of our study and to allow for subgroup analysis, we elected to enroll 200 patients. All statistical analyses were conducted using IBM-SPSS (version 29, Armonk NY, USA).

Descriptive analysis was performed for patients' demographics and the clinical characteristics of the study participants. Means and standard deviations were computed for continuous variables, and frequencies and percentages were calculated for categorical variables. Simple logistic regression was used to study the correlation between preoperative variables with the first attempt success rate. Also, simple logistic regression was used to study the association between preoperative variables, and the development of hypotension and hypoxemia during intubation. Variables with a P value < 0.25 were included in the multivariable logistic regression analysis. Multivariable logistic regression analysis was performed to identify the independent predictors of first attempt success rate, hypotension and hypoxemia during intubation, while adjusting for other preoperative variables. A P value < 0.05 was considered statistically significant. Multi-collinearity between covariates was assessed using Pearson's Correlation Coefficient. All models' fits were assessed using the Hosmer and Lemeshow test and using the C statistic, which is the area under the receiver operating characteristic curve.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective or emergent intubation on regular floors or ICU or COVID patients.
* Patients above 18 years of age.
* Intubation done by an anesthesia provider with at least 2 years of experience

Exclusion Criteria:

* Patients in the ED.
* Patients intubated by non-anesthesia providers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring elective or emergent endotracheal intubation
Sampling Method: Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
The success rate of endotracheal intubation at first attempt | During endotracheal intubation
  The success rate of endotracheal intubation at first attempt outside the OR

SECONDARY OUTCOMES:
Adverse events (Hypoxemia) | During the procedure
  Hypoxemia (SpO2 < 85%)
Adverse events (Hypotension) | During the procedure
  Hypotension (SBP < 80 mmHg)
Adverse events (cardiac arrest) | During the procedure
  Development of cardiac arrest
Total number of attempts | During the procedure
  Total number of attempts
Time to successful intubation | During the procedure
  Time to successful intubation in minutes
Equipment | During the procedure
  Type of equipments used (direct laryngoscopy/video laryngoscopy/awake fiberoptic)
Medications | During the procedure
  Type of medications used (Rocuronium, Midazolam, Propofol, vasoactive drugs)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Aouad-Maroun, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- AUBMC, Beirut, Lebanon